CLINICAL TRIAL: NCT01014468
Title: Comparative Study - Bevacizumab Versus Ranibizumab in Age Related Macular Degeneration
Brief Title: Bevacizumab Versus Ranibizumab in Age Related Macular Degeneration
Acronym: AxL-2009
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, Medical Doctor, Instituto de Olhos de Goiania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JJNJ - 8 - 2009
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Age Related Macular Degeneration
Keywords: ranibizumab; bevacizumab; AMD; Complications; Visual acuity; OCt; Age Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Intravitreal Injections; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Active Comparator): Intravitreal injection of Ranibizumab (3 monthly injection followed by monthly injections as long as required)
  Interventions: Drug: Ranibizumab (Intravitreal injection)
- Bevacizumab (Active Comparator): Intravitreal injection of Bevacizumab (3 monthly injection followed by monthly injections as long as required)
  Interventions: Drug: Bevacizumab (Intravitreal injection)

INTERVENTIONS:
Drug: Ranibizumab (Intravitreal injection) — Intravitreal injection of Ranibizumab 0.5 mg or Bevacizumab 1.25 mg (3 monthly injection followed by monthly
  Arms: Ranibizumab
Drug: Bevacizumab (Intravitreal injection) — Intravitreal injection of Ranibizumab 0.5 mg or Bevacizumab 1.25 mg (3 monthly injection followed by monthly
  Arms: Bevacizumab

SUMMARY:
To report the short term anatomic and visual acuity response after intravitreal injection of bevacizumab and ranibizumab in patients with choroidal neovascularization secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
We conducted a retrospective study of 500 eyes with choroidal neovascularization secondary to age-related macular degeneration who were treated with at least two (initial and one month after) intravitreal injection of 1.25 mg bevacizumab or 0.5 mg ranibizumab and had a follow-up of at least 3 months. Patients underwent Snellen visual acuity testing, optical coherence tomography (OCT) imaging and ophthalmoscopic examination at baseline and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Active primary or recurrent subfoveal lesion with CNV secondary to AMD

Exclusion Criteria:

* Prior treatment with any intravitreal drug in the study eye
* Prior treatment with verteporfin photodynamic therapy in the study eye
* Prior treatment with systemic bevacizumab
* Prior treatment with any intravitreal drug or verteporfin photodynamic therapy in the nonstudy eye within the 3 moths before the study entry
* Laser photocoagulation within 1 month before study entry in the study eye
* Previous participation in any clinical trial within 1 month before the entry of the study
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either of the two eye due to causes other than AMD such as histoplasmosis or pathological myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye that could either require medical or surgical intervention during the 12 month study period or that could contribute to a loss of best corrected visual acuity over the 12 months study period (e.g. diabetic retinopathy, cataract, uncontrolled glaucoma). The decision on exclusion is to be based on the opinion of the local principal investigator.
* Active intraocular inflammation
* Vitreous hemorrhage in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Vision change Anatomical changes (Regression of NVE, CNVM, reduction in macular thickness) Electrophysiological changes (ERG, VEP ) | 6 months

SECONDARY OUTCOMES:
Ocular side effects (infection, RD, IOP rise, cataract) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: João J Nassaralla, Jr, Study Chair — IOG and UnB
Locations (1):
- Instituto de Olhos de Goiânia, Goiânia, Goiás, Brazil